CLINICAL TRIAL: NCT00537797
Title: Limited Neck FDG-PET Imaging for Indeterminate Thyroid Nodules
Brief Title: Accuracy of FDG-PET Scanning to Diagnose Malignant Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-0757 / 201103045
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Thyroid Neoplasms
Keywords: Thyroid Neoplasms; Positron Emission Tomography; 18FDG
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 18-FDG-PET exam with SUV determination
  Thyroid operation to remove nodule
  Pathologic confirmation of nodule histology
  Determine sensitivity and specificity of FDG-PET, correlative studies
  Interventions: Other: FDG-PET Scan

INTERVENTIONS:
Other: FDG-PET Scan — Positron emission tomography with 18F-fluorodeoxyglucose

SUMMARY:
The main purpose of this study is to see how well FDG-PET scans can determine the malignancy of thyroid nodules that have already been tested (and come back positive) by fine needle aspiration.

DETAILED DESCRIPTION:
While FNA is a sensitive test for diagnosing thyroid tumors, it cannot differentiate benign from malignant follicular nodules and sometimes yields equivocal results due to inadequate sampling or indeterminate cytology. The standard of care for patients with equivocal or follicular histology is surgical removal of these nodules, most of which are benign in nature. FDG-PET, as evidenced by our prior experience and studies from other groups, may have application in discriminating benign from malignant disease in these patients with equivocal or follicular FNA results using standardized uptake value determination. We have demonstrated the feasibility and preliminary clinical utility of using limited neck FDG-PET exams in patients with indeterminate thyroid nodules in a pilot study. The purpose of this trial is to prospectively evaluate a larger series of patients with equivocal or follicular histology on FNA to more accurately define the sensitivity and specificity of FDG-PET for diagnostic imaging of these nodules. In addition, the utility of this modality in identifying metastatic foci in patients with thyroid cancer having follicular or equivocal histology on FNA will be assessed. If the sensitivity and specificity of this modality are determined to be high (≥95%) for diagnosing malignant nodules in these patients, many patients with benign disease may potentially benefit by avoiding unnecessary operations.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of a solitary thyroid nodule or a dominant nodule within multinodular disease, with fine needle aspiration demonstrating a follicular or indeterminate cytologic examination. If a core needle biopsy was performed instead of a fine needle aspiration, demonstrating follicular or indeterminate cytology, the patient is eligible if the biopsy procedure was felt to be minimally disruptive to the nodule architecture, based on a review by the PI or nuclear medicine investigator.
* Thyroid nodule must be palpable on physical examination or have a minimum size of 1 cm in diameter by ultrasonography, CT or MRI. The minimum size criterion was established to address the spatial resolution limitations of PET/CT imaging.
* Scheduled for surgical excision of thyroid nodules within 3 months of the date of the FDG-PET/CT scan.
* Ability to tolerate lying supine for a FDG-PET/CT examination.
* Age >/= 18 and </= 105 (This disease is rare in children and therefore the study will be limited to adults.)
* Willing to participate in all aspects of the study (patient may opt out of the tissue collection portion.)
* Patient must be euthyroid with a serum TSH or a free T4 level within the institutional upper and lower limits of normal, measured within 6 months of registration. NOTE: mild deviations from the institutional normal limits may be considered acceptable if the patient has achieved a clinically euthyroid state with medication at a stable dose for >3 months, and the TSH is considered to be at target by the patient's treating physician. In patients with hyperthyroidism requiring treatment, this euthyroid state may be achieved with administration of a thionamide such as propylthiouracil prior to FDG-PET/CT exam. Patients with hyperthyroid inflammatory conditions such as thyroiditis and toxic multinodular goiter often exhibit increased glucose uptake resulting in diffuse uptake of FDG which may obscure visualization of a thyroid tumor.
* If female, patient must have a negative pregnancy test at the time of registration, be post-menopausal (with no period in the last twelve months), have had a tubal ligation at least twelve months ago, or have had a hysterectomy.
* In patients with multinodular disease and a dominant nodule, the nuclear medicine physician responsible for FDG-PET/CT scan interpretation must determine whether the indeterminate nodule can be discriminated on FDG-PET/CT imaging prior to enrollment.
* A signed and dated written informed consent obtained from the patient or the patient's legally acceptable representative prior to study participation.

Exclusion Criteria:

* Patient has a fasting glucose level > 200 mg/dL at the time of the PET/CT scan
* Patient has had prior neck surgery or radiation that in the opinion of the investigator has disrupted tissue architecture of the thyroid
* Patient has evidence of infection localized to the neck in the 14 days prior to the FDG-PET/CCT scan
* Patient does not meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-08; Primary Completion 2011-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity and specificity of FDG-PET in identifying malignant thyroid nodules of follicular or indeterminate cytology. | Approximately 6 weeks after surgery
Estimate positive and negative predictive value of FDG-PET in identifying malignant thyroid nodules of follicular or indeterminate cytology. | Approximately 6 weeks after surgery
Estimate false positive rate and false negative rate of FDG-PET in identifying malignant thyroid nodules of follicular or indeterminate cytology. | Approximately 6 weeks after surgery

SECONDARY OUTCOMES:
Evaluate the sensitivity of the FDG-PET/CT imaging in localizing foci of metastatic disease within the neck in patients with thyroid malignancy identified as having follicular or equivocal histology by FNA | Approximately 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Moley, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - VAMC, St Louis, Missouri

REFERENCES:
- [Background] Lind P. Multi-tracer imaging of thyroid nodules: is there a role in the preoperative assessment of nodular goiter? Eur J Nucl Med. 1999 Aug;26(8):795-7. doi: 10.1007/s002590050450. No abstract available. PMID 10436189
- [Background] Jana S, Abdel-Dayem HM, Young I. Nuclear medicine and thyroid cancer. Eur J Nucl Med. 1999 Dec;26(12):1528-32. doi: 10.1007/s002590050490. No abstract available. PMID 10638402
- [Background] Mazzaferi, E., Radioiodine and other treatments and outcomes. Werner & Ingbar's the thyroid : a fundamental and clinical text ; editors, Lewis E. Braverman, Robert D. Utiger., 1996. 7th edn. Philadelphia: J.B. Lippincott-Raven: p. 922-943.
- [Background] Galloway RJ, Smallridge RC. Imaging in thyroid cancer. Endocrinol Metab Clin North Am. 1996 Mar;25(1):93-113. doi: 10.1016/s0889-8529(05)70314-5. PMID 8907682
- [Background] Wang W, Larson SM, Fazzari M, Tickoo SK, Kolbert K, Sgouros G, Yeung H, Macapinlac H, Rosai J, Robbins RJ. Prognostic value of [18F]fluorodeoxyglucose positron emission tomographic scanning in patients with thyroid cancer. J Clin Endocrinol Metab. 2000 Mar;85(3):1107-13. doi: 10.1210/jcem.85.3.6458. PMID 10720047
- [Background] Bloom AD, Adler LP, Shuck JM. Determination of malignancy of thyroid nodules with positron emission tomography. Surgery. 1993 Oct;114(4):728-34; discussion 734-5. PMID 8211687
- [Background] Bell RM. Thyroid carcinoma. Surg Clin North Am. 1986 Feb;66(1):13-30. doi: 10.1016/s0039-6109(16)43827-2. PMID 3511551
- [Background] Grant CS, Hay ID, Gough IR, McCarthy PM, Goellner JR. Long-term follow-up of patients with benign thyroid fine-needle aspiration cytologic diagnoses. Surgery. 1989 Dec;106(6):980-5; discussion 985-6. PMID 2588125
- [Background] Yousem DM, Scheff AM. Thyroid and parathyroid gland pathology. Role of imaging. Otolaryngol Clin North Am. 1995 Jun;28(3):621-49. PMID 7675472
- [Background] Goellner JR, Gharib H, Grant CS, Johnson DA. Fine needle aspiration cytology of the thyroid, 1980 to 1986. Acta Cytol. 1987 Sep-Oct;31(5):587-90. PMID 3673463
- [Background] Udelsman R, Westra WH, Donovan PI, Sohn TA, Cameron JL. Randomized prospective evaluation of frozen-section analysis for follicular neoplasms of the thyroid. Ann Surg. 2001 May;233(5):716-22. doi: 10.1097/00000658-200105000-00016. PMID 11323510
- [Background] Roach JC, Heller KS, Dubner S, Sznyter LA. The value of frozen section examinations in determining the extent of thyroid surgery in patients with indeterminate fine-needle aspiration cytology. Arch Otolaryngol Head Neck Surg. 2002 Mar;128(3):263-7. doi: 10.1001/archotol.128.3.263. PMID 11886341
- [Background] Strauss LG, Conti PS. The applications of PET in clinical oncology. J Nucl Med. 1991 Apr;32(4):623-48; discussion 649-50. PMID 2013803
- [Background] Rigo P, Paulus P, Kaschten BJ, Hustinx R, Bury T, Jerusalem G, Benoit T, Foidart-Willems J. Oncological applications of positron emission tomography with fluorine-18 fluorodeoxyglucose. Eur J Nucl Med. 1996 Dec;23(12):1641-74. doi: 10.1007/BF01249629. PMID 8929320
- [Background] Adler LP, Bloom AD. Positron emission tomography of thyroid masses. Thyroid. 1993 Fall;3(3):195-200. doi: 10.1089/thy.1993.3.195. PMID 8257858
- [Background] Grunwald F, Kalicke T, Feine U, Lietzenmayer R, Scheidhauer K, Dietlein M, Schober O, Lerch H, Brandt-Mainz K, Burchert W, Hiltermann G, Cremerius U, Biersack HJ. Fluorine-18 fluorodeoxyglucose positron emission tomography in thyroid cancer: results of a multicentre study. Eur J Nucl Med. 1999 Dec;26(12):1547-52. doi: 10.1007/s002590050493. PMID 10638405
- [Background] Feine U, Lietzenmayer R, Hanke JP, Held J, Wohrle H, Muller-Schauenburg W. Fluorine-18-FDG and iodine-131-iodide uptake in thyroid cancer. J Nucl Med. 1996 Sep;37(9):1468-72. PMID 8790195
- [Background] Cohen MS, Arslan N, Dehdashti F, Doherty GM, Lairmore TC, Brunt LM, Moley JF. Risk of malignancy in thyroid incidentalomas identified by fluorodeoxyglucose-positron emission tomography. Surgery. 2001 Dec;130(6):941-6. doi: 10.1067/msy.2001.118265. PMID 11742321
- [Background] Allal AS, Dulguerov P, Allaoua M, Haenggeli CA, El-Ghazi el A, Lehmann W, Slosman DO. Standardized uptake value of 2-[(18)F] fluoro-2-deoxy-D-glucose in predicting outcome in head and neck carcinomas treated by radiotherapy with or without chemotherapy. J Clin Oncol. 2002 Mar 1;20(5):1398-404. doi: 10.1200/JCO.2002.20.5.1398. PMID 11870185
- [Background] Yasuda S, Shohtsu A, Ide M, Takagi S, Takahashi W, Suzuki Y, Horiuchi M. Chronic thyroiditis: diffuse uptake of FDG at PET. Radiology. 1998 Jun;207(3):775-8. doi: 10.1148/radiology.207.3.9609903.
- [Background] Xu M, L.W., Cutler PD, Digby WM, Local threshold for segmented attenuation correction of PET imaging of the thorax. IEEE Trans Nuc Sci 1994. 41: p. 1532-7.
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu